CLINICAL TRIAL: NCT01755962
Title: Glycemic Load & Resistance Training on Endothelial Function & Insulin Sensitivity
Acronym: GET FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 546464
Record Dates: First submitted 2012-10-11; First posted 2012-12-24 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: 160 Participants Aged 18-35 Years and Obese (BMI ≥30) Open to Men and Women of All Ethnicity
Keywords: diet; obese; overweight; exercise; resistance training; nutrition; glycemic load; body composition; weight training; lifestyle
MeSH Terms: conditions — Obesity; Overweight; Motor Activity | interventions — Glycemic Load; Resistance Training

STUDY DESIGN:
Intervention Model Description: There are four intervention arms designed to compare two factors, glycemic load and resistance training. Arms consist of high glycemic diet, no exercise, high glycemic diet, resistance training; low glycemic diet, no exercise; low glycemic diet, resistance training.
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low Glycemic Load + Resistance Training (Experimental): 12-week intervention diet + resistance training (1 hour, 3 times per week)
  Interventions: Other: Glycemic Load; Other: Resistance Training
- High Glycemic Load + Resistance Training (Experimental): 12-week control diet + resistance training (1 hour, 3 times per week)
  Interventions: Other: Glycemic Load; Other: Resistance Training
- Low Glycemic Load (Experimental): 12-week intervention diet
  Interventions: Other: Glycemic Load
- High Glycemic Load (Other): 12-week control diet
  Interventions: Other: Glycemic Load

INTERVENTIONS:
Other: Glycemic Load
Other: Resistance Training
  Arms: High Glycemic Load + Resistance Training; Low Glycemic Load + Resistance Training

SUMMARY:
This project is prompted by the urgent public health need to identify novel strategies to prevent cardiovascular disease (CVD) and type 2 diabetes (T2D). The higher prevalence of CVD, T2D, and metabolic syndrome in obese individuals is a major healthcare concern. Therefore, finding optimal intervention strategies to combat these growing epidemics is imperative.

DETAILED DESCRIPTION:
At present, the extent to which dietary components can modify endothelial function, monocyte inflammation and glycemic variations is not well defined, although different carbohydrates are known to vary in their abilities to induce plasma glucose and insulin responses. Epidemiologic work suggests that high dietary glycemic load (GL) is associated with increased concentrations of inflammatory cytokines, endothelial dysfunction markers, and increased risk of T2D and coronary heart disease (CHD). We are examining using randomized control trials low vs. high-GL diet to determine if low-GL diets induce improvements in endothelial function or monocyte inflammation. Furthermore, resistance training is an alternate form of exercise from conventional aerobic training. Resistance Training has the potential to improve endothelial function or monocyte phenotype, but there is very little data in this area. We hypothesize that resistance training may augment the beneficial effects of a low-GL diet in improving metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 with BMI≥30 and/or your waist circumference ≥40 inches for males or ≥35 inches for females
* In good health as determined by the screening visit and review of medical history

Exclusion Criteria:

* Have a known heart arrhythmia and/or abnormalities found in electrocardiogram (ECG) reading or use of medications that influence CV function
* Have been in a weight loss or exercise program in the 6 months prior to participation
* Use tobacco products
* Have a syndrome or are prescribed medications that may influence body composition, insulin action, or CVD (e.g. PCOS, prednisone, methylphenidate, etc.)
* Have intolerance to lactose or gluten
* Pregnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2012-04; Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Endothelial function as determined by brachial artery FMD | 12 weeks

SECONDARY OUTCOMES:
monocyte inflammation | 12 weeks
Insulin Sensitivity by Oral Glucose Tolerance Test | 12 weeks
MAGE via Continuous Glucose Monitoring System | 12 weeks

OTHER OUTCOMES:
body composition (total fat mass, visceral fat, HFF, LBM) via DXA and MRI | 12 weeks
plasma and cellular biomarkers post pre and post 12 week intervention | 12 weeks
  Monocytes will be isolated from subject whole blood and will be phenotyped in 2 ways: 1) as pro- or anti-inflammatory based on flow-activated cell sorting (FACS) analysis of monocyte-specific markers TLR-4, CD14 and CD16.
  Serum-Stimulated Cell Culture. Subject serum will be incubated with L6 cells as we have previously performed in monocytes and adipocytes as well as endothelial cells 18, 130. Following 48 hr incubation, cellular insulin-stimulated glucose transport will be assayed as described 129 and conditioned medium assayed for myokine levels (ex. IL-15, 1L-6, etc).
  Fasting plasma (and conditioned media where appropriate) will be taken to determine a panel of adipokines and hormones (e.g. insulin, adiponectin, HSP-72, IL-4, IL-6, IL-10, MCP-1, CRP, 8-iso PGF2α) will be measured using the Millipore Multiplex assay kit or with specific ELISA kits
RNA/protein levels via muscle and fat tissue collection | 12 weeks
  Approximately 300 mg of muscle tissue from the superficial portion of the vastus lateralis and approximately 3-5 g of subcutaneous adipose tissue from the periumbilical portion of the abdomen will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Carpenter, PhD, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States